CLINICAL TRIAL: NCT00277940
Title: Neoaortic Elastic Properties After Aortic Arch Reconstruction
Brief Title: Aortic Arch Reconstruction
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Director Research, Children's Healthcare of Atlanta
Other Study IDs: 03-042
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: Pediatric; Cardiac; Neoaortic Elastic Properties; Aortic Arch Reconstruction
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Abnormalities of the aorta have been identified in patients who have undergone repair of coarctation of the aorta by various surgical techniques. These abnormalities are thought to contribute to ventricular hypertrophy, hypertension and exercise intolerance. Aortic arch reconstruction is performed for a variety of lesions besides simple coarctation of the aorta; these include hypoplastic left heart syndrome and its variants. In the latter group of patients extensive reconstruction is performed usually with a pulmonary homograft. We have previously shown that the neo-aortic dimensions and geometry are abnormal. The elastic properties of the neo-aorta, however, have not previously been described.

DETAILED DESCRIPTION:
In the present study we proposed to examine neo-aortic properties in a cohort of children with single ventricle heart defects who have undergone the bi-directional Glenn procedure (with or without Norwood palliation) and compare them to a cohort of patients with single ventricle who have had no aortic arch interventions. Patients in both groups typically undergo the Fontan operation between 18-48 months of age. After arrival to the operating suite and the placement of routine instrumentation, a transesophageal echocardiography (TEE) is routinely obtained. All data needed for this protocol is obtained during this TEE.

The stiffness of the aorta will be determined by calculating the pressure-strain elastic modulus (Ep) and the stiffness index beta (β). They are calculated from the formula Ep=[Ps-Pd]/[Ds-Dd/Dd] and β = [ln Ps/Pd[Ds-Dd]. Pressure-strain elastic modulus measurements have been utilized to measure the stiffness of the aorta and carotid arteries in both adults and children with a high reproducibility and low interobserver variability. The stiffness index beta has been proposed as a better measure of aortic stiffness because of its independence from measured blood pressure. The ability of a vessel to distend to store extra volume due to pressure effects is known as its compliance. A vessel with a higher compliance will be more "stretchy" and will therefore be more favorable to holding a greater volume of blood rather than storing a lot of pressure energy. Conversely, a vessel with a lower compliance will be less "stretchy" and therefore be more favorable to storing a lot of pressure energy rather than holding a greater volume of blood. Essentially, if two vessels are of equal size (cross-sectional flow area and volume), but one vessel has a lower compliance, then a 1 milliliter change in volume of the lower compliance (less stretchy) vessel will result in a greater pressure increase than a 1 milliliter change in volume of the higher compliance (more stretchy) vessel. Compliance will be assessed by the use of automatic border detection. This provides a continuous measure of the vessel cross-sectional area over time. Compliance is calculated by (Areamax-Areamean/mean blood pressure).

Blood pressure data will be recorded simultaneously with an arterial catheter that is used routinely during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Single ventricle congenital heart disease 1) palliated with bi-directional Glenn procedure after having the Norwood procedure (experimental group) or 2) palliated with the bi-directional Glenn without having the Norwood procedure as stage I palliation-i.e. Tricuspid Atresia, Pulmonary Atresia (control group)

Undergoing routine Fontan procedure

Exclusion Criteria:

* Semi-lunar valve insufficiency > trivial

Residual coarctation noted on routine pre-Fontan catheterization

Those who do not meet inclusion criteria

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: retro chart review
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States